CLINICAL TRIAL: NCT03548012
Title: Testing a Caregiver-led Intervention to Improve Support to Caregivers of Cancer Patients in Palliative Care at Home: a Stepped Wedge (Cluster) Randomized Controlled Trial
Brief Title: Improvement of Support to Caregivers of Cancer Patients in Basic Palliative Care at Home
Acronym: PiH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Danish Cancer Society (Other); Home care nursing in the Municipality of Gentofte (Unknown); Home care nursing in the Municipality of Gladsaxe (Unknown); Home care nursing in the Municipality of Haderslev (Unknown); Home care nursing in the Municipality of Holbæk (Unknown); Home care nursing in the Municipality of Odense (Unknown); Aalborg Municipality (Other); Home care nursing in the Municipality of Esbjerg (Unknown); Home care nursing in the Municipality of Hjørring (Unknown); Home care nursing in the Municipality of Næstved (Unknown); Home care nursing in the Municipality of Silkeborg (Unknown)
Responsible Party: Principal Investigator, Mogens Groenvold, Professor, DMSc, PhD, MD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R173-A11289-17-S51
Record Dates: First submitted 2018-05-22; First posted 2018-06-06 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Palliative Care
Keywords: Caregivers; Support Needs; Intervention; Randomised controlled trial
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: A stepped wedge cluster randomized controlled trial. All clusters (i.e., municipalities) will start as controls and will change to intervention at various times determined by randomization. In this way, all municipalities will contribute to control and intervention groups, thus accounting for variation between municipalities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Carer Support Needs Assessment Tool (CSNAT) intervention (Experimental): ('Standard' basic palliative care +) The Carer Support Needs Assessment Tool (CSNAT) intervention.
  Interventions: Behavioral: The Carer Support Needs Assessment Tool (CSNAT) intervention
- Control (No Intervention): ('Standard' basic palliative care). No intervention offered.

INTERVENTIONS:
Behavioral: The Carer Support Needs Assessment Tool (CSNAT) intervention — The CSNAT intervention is a caregiver-led approach where the caregiver first identifies his/her needs of support in the CSNAT, which consists of 14 support domains. Then the practitioner facilitates the intervention where the caregiver prioritizes which domains to discuss. In the conversation, the caregiver's domain priorities and subsequently identified support needs are discussed with the practitioner to agree on actions/solutions and a shared action plan. The intervention will be offered each caregiver twice: the first time between 0 and 13 days after enrollment, and the second time between 15 and 27 days after enrollment.
  Arms: The Carer Support Needs Assessment Tool (CSNAT) intervention

SUMMARY:
The aim of the project is to evaluate the use of the caregiver-led 'CSNAT intervention' to identify, prioritize and address support needs among caregivers of cancer patients who are starting in basic palliative care at home in Denmark

ELIGIBILITY:
Inclusion Criteria:

* The patient should have advanced cancer
* The caregiver and patient should be able to read and understand Danish
* The caregiver and patient should give written informed consent
* The patient should be newly referred to basic palliative care (BPC) by home nurses in the municipality.

Exclusion Criteria:

* The caregiver is viewed by the practitioners as being too distressed to be asked about participation
* The caregiver has a known cognitive impairment precluding participation (based on the practitioners' clinical judgement)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
Caregiver strain | Change from baseline (enrollment) to day 14
  Caregiver strain is measured by the subscale 'Caregiver Strain' in the Family Appraisal of Caregiving Questionnaire for Palliative Care (FACQ-PC). Subscale score range: 1-5. A higher score represents a worse outcome, i.e. more caregiver strain.

SECONDARY OUTCOMES:
Caregiver strain | Change from baseline (enrollment) to day 28
  Caregiver strain is measured by the subscale 'Caregiver Strain' in the Family Appraisal of Caregiving Questionnaire for Palliative Care (FACQ-PC). Subscale score range: 1-5. A higher score represents a worse outcome, i.e. more caregiver strain.
Positive caregiving appraisals | Change from baseline (enrollment) to day 14
  Positive caregiving appraisals is measured by the subscale 'Positive caregiving appraisals' in the Family Appraisal of Caregiving Questionnaire for Palliative Care (FACQ-PC). Subscale score range: 1-5. A higher score represents a better outcome, i.e. more positive caregiving appraisals.
Positive caregiving appraisals | Change from baseline (enrollment) to day 28
  Positive caregiving appraisals is measured by the subscale 'Positive caregiving appraisals' in the Family Appraisal of Caregiving Questionnaire for Palliative Care (FACQ-PC). Subscale score range: 1-5. A higher score represents a better outcome, i.e. more positive caregiving appraisals.
Caregiver distress | Change from baseline (enrollment) to day 14
  Caregiver distress is measured by the subscale 'Caregiver distress' in the Family Appraisal of Caregiving Questionnaire for Palliative Care (FACQ-PC). Subscale score range: 1-5. A higher score represents a worse outcome, i.e. more caregiver distress
Caregiver distress | Change from baseline (enrollment) to day 28
  Caregiver distress is measured by the subscale 'Caregiver distress' in the Family Appraisal of Caregiving Questionnaire for Palliative Care (FACQ-PC). Subscale score range: 1-5. A higher score represents a worse outcome, i.e. more caregiver distress
Satisfaction with attention from health care professionals | Change from baseline (enrollment) to day 14
  Measured by the subscale 'Lack of attention from health care professionals on the caregivers' wellbeing' in the Cancer Caregiving Tasks, Consequences and Needs Questionnaire (CaTCoN). Subscale score range: 0-100. A higher score represents a worse outcome, i.e. more lack of attention from health care professionals
Satisfaction with attention from health care professionals | Change from baseline (enrollment) to day 28
  Measured by the subscale 'Lack of attention from health care professionals on the caregivers' wellbeing' in the Cancer Caregiving Tasks, Consequences and Needs Questionnaire (CaTCoN). Subscale score range: 0-100. A higher score represents a worse outcome, i.e. more lack of attention from health care professionals
Satisfaction with communication with health care professionals | Change from baseline (enrollment) to day 14
  Measured by the subscale 'Problems with the quality of information from and communication with health care professionals' in the Cancer Caregiving Tasks, Consequences and Needs Questionnaire (CaTCoN). Subscale score range: 0-100. A higher score represents a worse outcome, i.e. more problems with the quality of information from and communication with health care professionals
Satisfaction with communication with health care professionals | Change from baseline (enrollment) to day 28
  Measured by the subscale 'Problems with the quality of information from and communication with health care professionals' in the Cancer Caregiving Tasks, Consequences and Needs Questionnaire (CaTCoN). Subscale score range: 0-100. A higher score represents a worse outcome, i.e. more problems with the quality of information from and communication with health care professionals
Satisfaction with information from health care professionals | Change from baseline (enrollment) to day 14
  Measured with selected items from the subscale 'Lack of information from health care professionals' in the Cancer Caregiving Tasks, Consequences and Needs Questionnaire (CaTCoN). Item/subscale score range: 0-100. A higher score represents a worse outcome, i.e. more lack of information from health care professionals
Satisfaction with information from health care professionals | Change from baseline (enrollment) to day 28
  Measured with selected items from the subscale 'Lack of information from health care professionals' in the Cancer Caregiving Tasks, Consequences and Needs Questionnaire (CaTCoN). Item/subscale score range: 0-100. A higher score represents a worse outcome, i.e. more lack of information from health care professionals
Caregiving workload | Change from baseline (enrollment) to day 14
  Measured with selected items from the subscale 'Caregiving workload' in the Cancer Caregiving Tasks, Consequences and Needs Questionnaire (CaTCoN). Item/subscale score range: 0-100. A higher score represents a worse outcome, i.e. more caregiving workload
Caregiving workload | Change from baseline (enrollment) to day 28
  Measured with selected items from the subscale 'Caregiving workload' in the Cancer Caregiving Tasks, Consequences and Needs Questionnaire (CaTCoN). Item/subscale score range: 0-100. A higher score represents a worse outcome, i.e. more caregiving workload
Caregiver involvement | Change from baseline (enrollment) to day 14
  Measured with item 12 in the Caregiving Tasks, Consequences and Needs Questionnaire (CaTCoN). Item score range: 0-100. A higher score represents a worse outcome, i.e. more caregiver dissatisfaction with involvement
Caregiver involvement | Change from baseline (enrollment) to day 28
  Measured with item 12 in the Caregiving Tasks, Consequences and Needs Questionnaire (CaTCoN). Item score range: 0-100. A higher score represents a worse outcome, i.e. more caregiver dissatisfaction with involvement
Help from health care professionals | Change from baseline (enrollment) to day 14
  Measured with two newly developed items which ask whether the health care professionals have talked with the caregiver about what burdens them, and whether the health care professionals have helped with these burdens. Item score range: 0-100. A higher score represents a worse outcome, i.e. less help from health care professionals
Help from health care professionals | Change from baseline (enrollment) to day 28
  Measured with two newly developed items which ask whether the health care professionals have talked with the caregiver about what burdens them, and whether the health care professionals have helped with these burdens. Item score range: 0-100. A higher score represents a worse outcome, i.e. less help from health care professionals
Quality of life | Change from baseline (enrollment) to day 14
  Measured by the two items assessing overall health and quality of life in the EORTC Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). Item score range: 0-100. A higher score represents a better outcome, i.e. better quality of life
Quality of life | Change from baseline (enrollment) to day 28
  Measured by the two items assessing overall health and quality of life in the EORTC Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). Item score range: 0-100. A higher score represents a better outcome, i.e. better quality of life
Emotional functioning | Change from baseline (enrollment) to day 14
  Measured by the four emotional functioning items in EORTC Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) supplemented with three selected items from the EORTC Computerized Adaptive Test (CAT) emotional functioning item bank. Item/subscale score range: 0-100. A higher score represents a better outcome, i.e. better emotional functioning
Emotional functioning | Change from baseline (enrollment) to day 28
  Measured by the four emotional functioning items in EORTC Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) supplemented with three selected items from the EORTC Computerized Adaptive Test (CAT) emotional functioning item bank. Item/subscale score range: 0-100. A higher score represents a better outcome, i.e. better emotional functioning
Fatigue | Change from baseline (enrollment) to day 14
  Measured by the three fatigue items in EORTC Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) supplemented with three selected items from the EORTC Computerized Adaptive Test (CAT) fatigue item bank. Item/subscale score range: 0-100. A higher score represents a worse outcome, i.e. more fatigue
Fatigue | Change from baseline (enrollment) to day 28
  Measured by the three fatigue items in EORTC Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) supplemented with three selected items from the EORTC Computerized Adaptive Test (CAT) fatigue item bank. Item/subscale score range: 0-100. A higher score represents a worse outcome, i.e. more fatigue
Positive emotional functioning | Change from baseline (enrollment) to day 14
  Measured by five positively formulated items concerning emotional functioning which were excluded from the EORTC Computerized Adaptive Test (CAT) emotional functioning bank during the development of the item bank. Item score range: 0-100. A higher score represents a better outcome, i.e. more positive emotional functioning
Positive emotional functioning | Change from baseline (enrollment) to day 28
  Measured by five positively formulated items concerning emotional functioning which were excluded from the EORTC Computerized Adaptive Test (CAT) emotional functioning bank during the development of the item bank. Item score range: 0-100. A higher score represents a better outcome, i.e. more positive emotional functioning
Caregiver grief | Measured six months after the patient's death
  Measured by the Prolonged Grief Scale-13 (PG-13). Symptom subscale score range: 9-45. A higher score represents a worse outcome, i.e. higher level of prolonged grief symptoms
Acute hospitalizations | Change from baseline (enrollment) to day 14
  Number of acute patient hospitalizations
Acute hospitalizations | Change from baseline (enrollment) to day 28
  Number of acute patient hospitalizations
Hospice referrals (for in-patient care) | Change from baseline (enrollment) to day 14
  Number of patients referred to hospice in-patient care
Hospice referrals (for in-patient care) | Change from baseline (enrollment) to day 28
  Number of patients referred to hospice in-patient care
Survival time | From enrollment to up to six months after the project recruitment period has closed
  Number of days the patient lives
Place of death | From enrollment to up to six months after the project recruitment period has closed
  The place in which the patient dies

CONTACTS AND LOCATIONS:
Overall Officials: Mogens Grønvold, DMSc PhD MD, Principal Investigator — Bispebjerg Hospital
Locations (10):
- Denmark (10):
  - Aalborg Home Nursing, Aalborg
  - Esbjerg Home Nursing, Esbjerg
  - Gentofte Home Nursing, Gentofte Municipality
  - Gladsaxe Home Nursing, Gladsaxe
  - Haderslev Home Nursing, Haderslev
  - Hjørring Home Nursing, Hjørring
  - Holbæk Home Nursing, Holbæk
  - Næstved Home Nursing, Næstved
  - Odense Home Nursing, Odense
  - Silkeborg Home Nursing, Silkeborg

IPD SHARING:
Plan to Share IPD: No